CLINICAL TRIAL: NCT03428074
Title: A Multi-centre Real-world Non-interventional Observational Study to Compare Effectiveness and Safety of the Minimally Invasive Surgeries of Ivor-Lewis and Mckeown in Chinese Patients With IA-IIIB Esophageal Cancer
Brief Title: A Observational Study to Compare Effectiveness and Safety of the Surgeries in Patients With Esophageal Cancer
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Yang Liu, Professor, Chinese PLA General Hospital
Other Study IDs: 301-EC-01
Record Dates: First submitted 2018-02-05; First posted 2018-02-09 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Esophageal Cancer
Keywords: Chinese, esophageal cancer, surgeries of Ivor-Lewis/Mckeown
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with the surgery of Ivor-Lewis: Pathologically diagnosed IA-IIIB patients with esophageal cancer who received minimally invasive surgery of Ivor-Lewis
  Interventions: Procedure: Surgeries
- Patients with the surgery of Mckeown: Pathologically diagnosed IA-IIIB patients with esophageal cancer who received minimally invasive surgery of Mckeown
  Interventions: Procedure: Surgeries

INTERVENTIONS:
Procedure: Surgeries — Minimally invasive surgeries of Ivor-Lewis and Mckeown

SUMMARY:
The study was designed to compare effectiveness and safety of the surgeries of Ivor-Lewis and Mckeown in patients with esophageal cancer

DETAILED DESCRIPTION:
The trial is a multi-centre real-world non-interventional observational study. The study was designed to compare effectiveness and safety of the minimally invasive surgeries of Ivor-Lewis and Mckeown in the Chinese patients with IA-IIIB esophageal cancer via a retrospectively review method based on the study data on patient demographic/tumor biological characteristics and clinical treatments.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed middle and lower thoracic IA-IIIB esophageal cancer after surgeries;
* Patients who received minimally invasive radical dissections of Ivor-Lewis and Mckeown;
* Patients who received tubular gastroesophageal reconstruction;

Exclusion Criteria:

* Patients complicated with arrhythmia, or serious disfunctions of heart, lung, liver, and kidney before surgeries;
* Patients with second primary tumors;
* Patients who received abdominal or thoracic surgeries;
* Patients who received gastrostomy or nesteostomy before surgeries;
* Patients with suspected cervical lymph metastases (in the subgroup of the patients who received the surgery of Mckeown)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pathogically diagnosed IA-IIIB patients with esophageal cancer who received the surgeries of Ivor-Lewis and Mckeown
Sampling Method: Non-Probability Sample
Enrollment: 1862 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Overall survivals in patients with esophageal cancer who received surgeries | 2010 - 2017
  Overall survivals in patients with esophageal cancer who received surgeries categorised by tumor biological characteristics

SECONDARY OUTCOMES:
Death rates within 30 days after surgeries | 2010 - 2017
  Death rates within 30 days after surgeries categorised by tumor biological characteristics

OTHER OUTCOMES:
Incidence of complications after surgeries | 2010 - 2017
  Incidence of complications after surgeries categorised by tumor biological characteristics
Incision R0 rates | 2010 - 2017
  Incision R0 rates categorised by tumor biological characteristics
Percentages of patients who received lymphadenectomy | 2010 - 2017
  Percentages of patients who received lymphadenectomy categorised by tumor biological characteristics
Extents of lymph metastases | 2010 - 2017
  Extents of lymph metastases categorised by tumor biological characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Yang Liu, PhD, Principal Investigator — Chinese PLA General Hospital
Locations (9):
- China (9):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Henan cancer hospital, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Huazhong Technology Hospital, Wuhan, Hubei
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Xi'an Tangdu Hospital, Xi'an, Shaanxi
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Huaxi Hospital Affiliated to Sichuan University, Chengdu, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - First Hospital Affiliated to Medical College, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang T, Hou X, Li Y, Fu X, Liu L, Xu L, Liu Y. Effectiveness and safety of minimally invasive Ivor Lewis and McKeown oesophagectomy in Chinese patients with stage IA-IIIB oesophageal squamous cell cancer: a multicentre, non-interventional and observational study. Interact Cardiovasc Thorac Surg. 2020 Jun 1;30(6):812-819. doi: 10.1093/icvts/ivaa038. PMID 32285107